CLINICAL TRIAL: NCT05812534
Title: Phase II Study of Cadonilimab Combined With Bevacizumab and Chemotherapy for Advanced Nonsquamous Non-small Cell Lung Cancer Patients With Untreated Brain Metastases
Brief Title: Study of Cadonilimab Combined With Bevacizumab and Chemotherapy for Advanced Nonsquamous Non-small Cell Lung Cancer Patients With Untreated Brain Metastases
Acronym: CBC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital of Nanchang University (Other)
Collaborators: Hunan Cancer Hospital (Other); Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT-I-2022-050
Record Dates: First submitted 2023-02-27; First posted 2023-04-13 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Non Small Cell Lung Cancer; Brain Metastases
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental group (Experimental): Subjects who met the study population conditions were treated with Cadonilimab 10mg/kg + bevacizumab 7.5 mg/kg + carboplatin (AUC 5) + pemetrexed 500mg/m2. Every 3 weeks is a cycle, with a total of 4-6 cycles (the number of chemotherapy cycles is determined by the researchers). Cadonilimab 10mg/kg, bevacizumab 7.5 mg/kg and pemetrexed 500mg/m2 were then maintained until disease progression, intolerable toxicity or other causes specified in the regimen occurred. When the subject first has imaging disease progression, if the researcher judges that it is clinically beneficial and tolerant to the test drug, he will be allowed to continue treatment.
  Interventions: Drug: Cadonilimab

INTERVENTIONS:
Drug: Cadonilimab — Subjects who met the study population conditions were treated with Cadonilimab 10mg/kg + bevacizumab 7.5 mg/kg + carboplatin (AUC 5) + pemetrexed 500mg/m2. Every 3 weeks is a cycle, with a total of 4-6 cycles (the number of chemotherapy cycles is determined by the researchers). Cadonilimab 10mg/kg, bevacizumab 7.5 mg/kg and pemetrexed 500mg/m2 were then maintained until disease progression, intolerable toxicity or other causes specified in the regimen occurred. When the subject first has imaging disease progression, if the researcher judges that it is clinically beneficial and tolerant to the test drug, he will be allowed to continue treatment.

SUMMARY:
The purpose of this study was to investigate the efficacy and safety of Cadonilimab combined with bevacizumab and chemotherapy for advanced non-squamous NSCLC with untreated brain metastases. Cadonilimab is a bispecific antibody (BsAb), which can bind PD-1 and CTLA-4 at the same time with high affinity. It is a new tumor immunotherapy drug with tetravalent structure and short half-life. It has shown less toxicity than anti-PD-1 and anti-CTLA-4 antibodies in monkey toxicity studies. These characteristics make the application of Cadonilimab in tumor subjects may have better efficacy and safety.

AK104-207 is an open, multicenter, phase Ib/II clinical study, which aims to evaluate the effectiveness and safety of Cadonilimab combined with chemotherapy as the first-line treatment for locally advanced or metastatic non-small cell lung cancer that cannot be operated and cannot receive radical concurrent/sequential radiotherapy and chemotherapy. As of August 1, 2022, 19 subjects who can evaluate non-squamous NSCLC (cohort B), ORR is 63.2%, DCR is 100%, median PFS is 13.34 months (7.36, NE), median OS is not reached, and 12-month OS rate is 76.0% (95% CI 48.0-90.3). In PD-L1 positive patients (n=9), ORR was 55.6% and DCR was 100%. In PD-L1 negative patients (n=7), ORR was 85.7% and DCR was 100%.

In view of the early curative effect of Cadonilimab in NSCLC single drug or combination therapy and the encouraging research results of PD-1 inhibitor combined with CTLA-4 double immune combination therapy, it is expected that Cadonilimab combined with bevacizumab and chemotherapy will achieve good curative effect in NSCLC patients with brain metastasis.

DETAILED DESCRIPTION:
Study Name:

Phase II study of Cadonilimab combined with bevacizumab and chemotherapy for advanced nonsquamous non-small cell lung cancer patients with untreated brain metastases Purpose of research MAIN OBJECTIVE: Total response rate (ORR) Secondary purposes: progression-free survival (PFS), intracranial PFS (iPFS), overall survival (OS), Quality of Life (QoL) and safety Exploratory Objective: To explore the potential evolutionary mechanism of brain metastasis of lung cancer and the difference of immune microenvironment between primary focus and metastatic focus.

Design type: Intervention research Subjects: Non-squamous NSCLC in advanced stage of untreated brain metastasis Sample size: 36 cases Statistical analysis method: This cohort was a one-arm test, using Simon-Minimax two-stage design, assuming that the ORR rate was 20% under the ineffective hypothesis and 40% under the hypothesis that the drug was considered effective. The degree of assurance is 0.8, the test level α is set to 0.05, and the sample size estimation result is a total sample of 33 cases. Eighteen subjects who meet the admission criteria are planned to be enrolled first. If 4 patients have CR or PR, they will continue to be enrolled until 33 patients are reached. Only when more than 10 patients in the total sample reach CR or PR can the study reach the main endpoint. Considering the shedding rate of 10%, the sample size of this study is estimated to be 36 cases. Data were collected from the first day of treatment to the death of the patient or the last follow-up. All rate estimates were evaluated by Kaplan-Meier model (SPSS, version 25.0). Univariate analysis and multivariate analysis of Cox regression model were used to analyze the related factors of prognosis. long-rank test was used to compare the difference of observation endpoint. P < 0.05 was statistically significant.

Screening period: Subjects will complete screening evaluation within 28 days before the first medication to determine whether they meet the research conditions. During the screening period, the peripheral blood of the subjects should be collected.

Treatment period: The subjects who met the conditions of the study population were treated with Cadonilimab 10mg/kg + bevacizumab 7.5 mg/kg + carboplatin (AUC 5) + pemetrexed 500mg/m2. Every 3 weeks is a cycle, with a total of 4-6 cycles (the number of chemotherapy cycles is determined by the researchers). Cadonilimab 10mg/kg, bevacizumab 7.5 mg/kg and pemetrexed 500mg/m2 were then maintained until disease progression, intolerable toxicity or other causes specified in the regimen occurred. When the subject first has imaging disease progression, if the researcher judges that it is clinically beneficial and tolerant to the test drug, he will be allowed to continue treatment.

During the treatment, the researchers evaluated the curative effect according to RECIST 1.1 standard. ORR evaluated by researchers was used as the main curative effect index. Subjects were evaluated for tumor every 6 weeks (7 days) within 54 weeks after enrollment, and every 12 weeks (7 days) after enrollment. Subjects who stop taking drugs for non-disease progression reasons will continue to follow up their disease status until the subjects start other anti-tumor treatment, disease progression, withdrawal of consent, death or end of study, whichever occurs first.

During the treatment, researchers will collect a series of blood samples for pharmacokinetics, immunogenicity and exploratory research and analysis.

Adverse events (AE) of each subject will be collected until 30 days after the last administration or new anti-tumor treatment will be started, whichever occurs first. Serious adverse events (SAE) will be collected until 90 days after the last administration or new anti-tumor treatment will be started, whichever occurs first. Immune-related AE (irAE) will be collected until 90 days after the last administration or new anti-tumor therapy will be started, whichever occurs first. Survival assessment was performed every 3 months after the last dose to obtain survival information and collect information on subsequent anti-tumor treatment after termination of study treatment.

ELIGIBILITY:
Inclusion Criteria:

* The patient was over 18 years old.
* The Eastern Cooperative Oncology Group Performance Status score ranged from 0 to 1.
* Patients with asymptomatic brain metastases confirmed by histology or cytology as EGFR and ALK negative stage IV non-squamous NSCLC who have not received any chemotherapy or brain radiotherapy before.
* Patients with non-metastatic diseases who have received neoadjuvant chemotherapy, adjuvant chemotherapy or radiotherapy must experience a no-treatment interval of at least 6 months since the last chemotherapy and/or radiotherapy.
* Steroid therapy (dexamethasone) is allowed. When dexamethasone ≤ 4mg once a day, patients who are still asymptomatic or less symptomatic after 2 weeks of steroid use will be eligible.
* Extracranial measurable lesions assessed by CT (RECIST 1.1 standard), Intracranial measurable lesions (RANO-BM standard or brain MRI).
* Formalin-fixed paraffin embedded blocks (cell wax blocks are acceptable if no tumor biopsy is available) containing tumor tissue or 10 unstained slides can be obtained.
* Adequate hematopoiesis and liver and kidney function: ANC ≥ 1,500 cells/μ L, lymphocyte count ≥ 500 cells/μ L, platelet count ≥ 100,000 cells μ L, hemoglobin ≥ 9.0 g/dL (blood transfusion allowed); INR or aPTT ≤ 1.5 x upper normal limit (ULN); Patients receiving therapeutic anticoagulant therapy should use stable doses of ALT, AST and/or ALP ≤ 2.5 x ULN, except for the following (ALT and/or AST ≤ 5 x ULN in patients with known liver metastasis; ALP ≤ 5 x ULN in patients with known bone metastasis; Serum bilirubin ≤ 1.5 x ULN; Serum bilirubin ≤ 3 x ULN in patients with known Gilbert disease). Creatinine clearance rate (CRCL) ≥ 45 mL/min (based on standard Cockcroft and Gault formulas).
* For fertile women: agree to abstinence or use non-hormonal contraceptive methods during treatment and for 3 months after treatment in the last study. A woman is considered to have fertility potential if she is in the post-menarche state, has not reached the post-menopausal state (amenorrhea for 12 consecutive months, with no definite cause other than menopause) and has not undergone surgical sterilization (ovariectomy and/or uterus removal).
* For men: agree to keep abstinence or use condoms, and agree not to donate sperm. For fertile female partners or pregnant female partners, men must keep abstinence or use condoms during treatment and for three months after the last study treatment to avoid exposing embryos. In the meantime, men must avoid donating sperm.
* Sign the informed consent form.

Exclusion Criteria:

* History of other malignant tumors within 3 years before screening, except properly treated cervical carcinoma in situ, non-melanoma skin cancer or stage I uterine cancer.
* Patients with EGFR mutations or ALK fusion will be excluded.
* Metastasis of pia mater, brain stem, midbrain, pons and medulla or metastasis leading to obstructive hydrocephalus.
* Patients with neurological symptoms, including those receiving > 4mg dexamethasone, will not be eligible for inclusion in this study.
* Spinal or hemorrhagic metastases will be excluded.
* Surgical treatment of brain or spinal lesions within 14 days before.
* The previous systemic treatment or neoadjuvant or adjuvant chemotherapy before admission was less than 6 months.
* With clinically significant complications affecting platinum chemotherapy administration.
* Autoimmune history, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener granuloma, Sjogren's syndrome, Guillain-Barre syndrome, multiple sclerosis, vasculitis or glomerulonephritis. Exceptions to the following：①Patients with a history of autoimmune-associated hypothyroidism and taking a stable dose of thyroid replacement hormone are eligible for this study.

  ②Patients with controlled type 1 diabetes who received a steady dose of insulin were eligible for this study.

  ③Patients with eczema, psoriasis, chronic lichen simplex, or vitiligo with only dermatological manifestations (e.g. psoriatic arthritis patients will be excluded) provided they meet the following conditions: the rash covers less than 10% of the body surface area, the disease is well controlled at baseline, only inefficient topical steroids are required, and there is no acute attack in the past 12 months.
* History of idiopathic pulmonary fibrosis, drug-induced pneumonia or active radiation pneumonia in radiation field.
* Previous treatment was with immune checkpoint inhibitors or CD137 and OX-40 agonists.
* Receive research treatment within 28 days before starting the study drug, and screen for hepatitis C virus (HCV) antibody or hepatitis B surface antigen (HBsAg). Patients with previous or cured hepatitis B virus (HBV) infection (HBcAb positive but no HBsAg) are eligible regardless of their HBV DNA negative. Patients with positive HCV antibody are eligible regardless of whether HCV RNA is negative or not.
* Active tuberculosis or HIV infection.
* Abuse of drugs or alcohol within 12 months before screening.
* Any serious medical condition or abnormality in clinical laboratory examination prevents patients from safely participating in and completing the study according to the judgment of the researcher.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
overall response rate | 6 weeks
  The proportion of the total number of patients with complete response and partial response to the total number of evaluable cases.

SECONDARY OUTCOMES:
Intracranial Progress Free Survival rate | 24 months
  It is the time from clinical discovery of brain metastasis to the first intracranial progression or death.
Progress Free Survival rate | 24 months
  The period from the beginning of clinical study to the progression or death of the patient.
overall survival | 24 months
  The period from the beginning of clinical study to the death of the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Anwen Liu, PhD, Principal Investigator — Second Affiliated Hospital of Nanchang University

IPD SHARING:
Plan to Share IPD: Undecided